CLINICAL TRIAL: NCT01184859
Title: A Multi-centre, Double-blind, Randomised, Placebo-controlled, Parallel-group, Comparative Trial to Investigate the Dose-Response of 4 Different Dose Levels of Minirin Melt and Placebo in Water-loaded Male and Female Japanese Nocturia Patients (Single Dose), and to Study the Efficacy of 4 Different Dose Levels of Minirin Melt and Placebo After 28 Days of Dosing (Multiple Doses)
Brief Title: Comparative Trial to Investigate the Dose-Response of 4 Different Dose Levels of Minirin Melt and Placebo
Acronym: NOC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FE992026 CS36
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Results first posted 2012-05-25 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-04

CONDITIONS: Nocturia
Keywords: nocturia; bladder function
MeSH Terms: conditions — Nocturia | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Desmopressin 10µg (Experimental): Study period 1: single dose of desmopressin 10µg. Study period 2: daily doses of desmopressin 10µg taken before bedtime for 28 days.
  Interventions: Drug: Desmopressin
- Desmopressin 25µg (Experimental): Study period 1: single dose of desmopressin 25µg. Study period 2: daily doses of desmopressin 25µg taken before bedtime for 28 days.
  Interventions: Drug: Desmopressin
- Desmopressin 50µg (Experimental): Study period 1: single dose of desmopressin 50µg. Study period 2: daily doses of desmopressin 50µg taken before bedtime for 28 days.
  Interventions: Drug: Desmopressin
- Desmopressin 100µg (Experimental): Study period 1: single dose of desmopressin 100µg. Study period 2: daily doses of desmopressin 100µg taken before bedtime for 28 days.
  Interventions: Drug: Desmopressin
- Placebo (Placebo Comparator): Study period 1: single dose of placebo. Study period 2: daily doses of placebo taken before bedtime for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Desmopressin — Desmopressin oral lyophilisate melt tablet, in either the 10, 25, 50, or 100 μg dosage, for sublingual administration
  Other Names: FE992026; Minirin Melt
  Arms: Desmopressin 100µg; Desmopressin 10µg; Desmopressin 25µg; Desmopressin 50µg
Drug: Placebo — Placebo melt tablet for sublingual administration
  Arms: Placebo

SUMMARY:
This is a multi-centre, randomised, placebo-controlled, double-blind, parallel-group comparative trial to be conducted in nocturia patients. The trial is designed to characterize the dose-response relationship of Minirin (desmopressin) Melt in order to establish correct dose recommendations in the target patient population. In particular, the trial is designed to link the duration of action to the clinical endpoint. Furthermore, the trial is designed to describe the safety of four different dose levels of desmopressin.

ELIGIBILITY:
Inclusion Criteria:

* Given written informed consent prior to any trial-related activity is performed
* Aged 55-75 years
* Mean number of nocturnal voids of at least two per night
* Reached post-menopause (applicable to females only)

Exclusion Criteria:

* Evidence of bladder outlet obstruction (BOO); or a urine flow of less than 5 mL/s (applicable to males only)
* A surgical treatment for BOO or prostatic hyperplasia within the past 6 months (applicable to males only)
* Showing symptoms of any of the following diseases and having a mean number of nocturnal voids exceeding four per night: Benign prostatic hyperplasia, overactive bladder, interstitial cystitis, severe stress urinary incontinence
* Psychosomatic or habitual polydipsia
* Urinary retention; or a post void residual volume in excess of 150 mL
* A history or complication of urologic malignancy (e.g. bladder cancer or prostate cancer)
* Complication of genito-urinary pathology (e.g. infection, stone, or neoplasia)
* Complication of neurogenic detrusor activity
* Complication or suspicion of heart failure
* Uncontrolled hypertension
* Uncontrolled diabetes mellitus
* Complication of hepatobiliary disease
* Abnormal serum creatinine level
* Complication of hyponatraemia, or serum sodium level <135 mEq/L
* Central or nephrogenic diabetes insipidus (CDI or NDI)
* Syndrome of inappropriate antidiuretic hormone (SIADH)
* Obstructive sleep apnea
* Alcohol dependency or drug abuse
* A job or lifestyle that may interfere with regular night-time sleep
* Previous desmopressin treatment
* Treatment with another investigational product within the past 3 months
* A need for treatment with a prohibited concomitant drug for a complication or other problem
* A mental condition, the lack of decision-making ability, dementia or a speech handicap
* Any other reason that the Investigator believes inappropriate

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (36):
- Japan (36):
  - Japanese Red Cross Nagoya Daiichi Hospital, Nagoya, Aichi-ken
  - National Center for Geriatrics and Gerontology, Ōbu, Aichi-ken
  - Kokuho Asahi Central Hospital, Asahi, Chiba
  - University of Fukui Hospital, Yoshida, Fukui
  - Takayama Hospital, Chikushino-shi, Fukuoka
  - Harasanshin Hospital, Fukuoka, Fukuoka
  - Saku Hospital, Fukuoka, Fukuoka
  - Southwest Urological Clinic, Fukuoka, Fukuoka
  - Yakuin Urogenital Hospital, Fukuoka, Fukuoka
  - Houshikai Group Kano Hospital, Koga, Fukuoka
  - St. Mary's Hospital, Kurume, Fukuoka
  - Fukushima Red Cross Hospital, Fukushima, Fukushima
  - Ohara General Hospital, Fukushima, Fukushima
  - Saiseikai Fukushima General Hospital, Fukushima, Fukushima
  - Jyusendo General Hospital, Kōriyama, Fukushima
  - Social Insurance Nihonmatsu Hospital, Nihommatsu, Fukushima
  - Takayama Clinic, Awagi, Hyōgo
  - National Hospital Organization Kobe Medical Center, Kobe, Hyōgo
  - Japanese Red Cross Mito Hospital, Mito, Ibaraki
  - Jigenji Kubo Clinic, Kagoshima, Kagoshima-ken
  - Kawahara Hinyoukika, Kagoshima, Kagoshima-ken
  - Yagi Clinic, Kagoshima, Kagoshima-ken
  - Yokohama Shin-midori General Hospital, Yokohama, Kanagawa
  - Kumamoto Rosai Hospital, Yatsushiro, Kumamoto
  - Rakusai Newtown Hospital, Kyoto, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Shinshu University Hospital, Matsumoto, Nagano
  - Suzuki Urological Clinic, Nagano, Nagano
  - Senbokufujii Hospital, Sakai, Osaka
  - Nanri Urological Clinic, Saga, Saga-ken
  - Kasukabe Chuo General Hospital, Kasukabe, Saitama
  - Hamamatsu University School of Medicine University Hospital, Hamamatsu, Shizuoka
  - Tokyo Women's Medical University Medical Center East, Arakawa City, Tokyo
  - Koganeibashi Sakura Clinic, Koganei, Tokyo
  - Kunitachi Sakura Hospital, Kunitachi, Tokyo
  - University of Yamanashi Hospital, Chūō, Yamanashi

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 139 patients randomized and 116 treated. Withdrawals during the screening period were due to urine production did not meet >0.12 mL/kg/min within 2 hours of dosing (22 patients) and violation of inclusion/exclusion criteria (1 patient).
Period: Period 1: Single Dose
Arm/Group | Placebo | Desmopressin 10µg | Desmopressin 25µg | Desmopressin 50µg | Desmopressin 100µg
Started | 23 | 25 | 22 | 22 | 24
Full Analysis Set (FAS) | 23 | 23 (2 participants disqualified due to no post-baseline primary efficacy data, and/or 'other'.) | 22 | 21 (1 participant disqualified due to major entry criteria violation) | 24
Per Protocol (PP) | 23 | 23 | 22 | 21 | 23 (1 additional participant disqualified due to 'other'.)
Completed | 23 | 23 | 22 | 22 | 23
Not Completed | 0 | 2 | 0 | 0 | 1
Not completed — Insufficient urine production | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Period: Washout Period
Arm/Group | Placebo | Desmopressin 10µg | Desmopressin 25µg | Desmopressin 50µg | Desmopressin 100µg
Started | 23 | 23 | 22 | 22 | 23
Completed | 23 | 23 | 22 | 22 | 23
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 2: Daily Dose for 28 Days
Arm/Group | Placebo | Desmopressin 10µg | Desmopressin 25µg | Desmopressin 50µg | Desmopressin 100µg
Started | 23 | 23 | 22 | 22 | 23
Completed | 22 | 23 | 22 | 22 | 22
Not Completed | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Desmopressin 10µg | Desmopressin 25µg | Desmopressin 50µg | Desmopressin 100µg | Total
Number analyzed (Participants) | 23 | 23 | 22 | 21 | 24 | 113
Age Continuous [Mean (Standard Deviation); unit: years] — FAS population is used for the Baseline Measures
  years | 64.3 (6.4) | 67.0 (5.6) | 65.5 (6.0) | 64.9 (7.1) | 65.3 (5.6) | 65.4 (6.1)
Age, Customized [Number; unit: participants]
  >=55 and <65 years | 12 | 8 | 10 | 10 | 12 | 52
  >=65 and <76 years | 11 | 15 | 12 | 11 | 12 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 11 | 11 | 12 | 58
  Male | 11 | 11 | 11 | 10 | 12 | 55
Number of Nocturnal Voids [Mean (Standard Deviation); unit: nocturnal voids] | 2.16 (0.26) | 2.43 (0.51) | 2.45 (0.45) | 2.29 (0.44) | 2.26 (0.38) | 2.32 (0.42)
Number of Daytime Voids [Mean (Standard Deviation); unit: daytime voids] | 7.67 (1.48) | 7.97 (1.91) | 8.70 (1.53) | 8.67 (1.99) | 8.33 (1.65) | 8.26 (1.74)
Number of 24-hour Voids [Mean (Standard Deviation); unit: voids] | 9.83 (1.52) | 10.41 (1.94) | 11.15 (1.79) | 10.95 (2.12) | 10.60 (1.60) | 10.58 (1.83)
Nocturnal Urine Volume [Mean (Standard Deviation); unit: mL] | 634.78 (210.54) | 568.55 (227.40) | 613.06 (182.47) | 635.87 (211.53) | 631.78 (175.02) | 616.64 (200.13)
24-Hour Urine Volume [Mean (Standard Deviation); unit: mL] | 1742.32 (344.99) | 1632.17 (454.75) | 1881.67 (399.42) | 1848.32 (497.96) | 1785.65 (404.67) | 1775.93 (423.67)

OUTCOME MEASURES:

1. Primary Outcome: Duration of Action Defined as the Time With Urine Osmolality Above 200 mOsm/kg - Period 1
Description: Participants were water-loaded to suppress the endogenous release of vasopressin, thus all antidiuretic activity was generated by desmopressin only. Water-loading was initiated 2 hours before dosing on Day 1. Urine volume was registered and samples for osmolality check were collected every 30 minutes as long as there was an antidiuretic action defined as a urine production <0.12 mL/kg/min. The hydration should have lasted until end of action, defined as when the urine production returned to >0.12 mL/kg/min, but no longer than 12 hours.
Time Frame: Day 1
Population: Per protocol population, consisting of treated participants without major protocol violations and with >=80% treatment compliance.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | Desmopressin 10µg | Desmopressin 25µg | Desmopressin 50µg | Desmopressin 100µg
Number analyzed (Participants) | 23 | 23 | 22 | 21 | 21
hours | 0.00 (0.00) | 0.09 (0.32) | 2.00 (3.56) | 3.45 (2.88) | 5.74 (2.99)
Statistical Analysis 1: Comparison: Placebo vs Desmopressin 10µg; Test type: Superiority or Other; p = 0.211, t-test, 2 sided — The p-value was not adjusted for multiplicity, because this study was not a confirmatory trial. A priori threshold for statistical significance is 0.05
Statistical Analysis 2: Comparison: Placebo vs Desmopressin 25µg; Test type: Superiority or Other; p = 0.010, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Desmopressin 50µg; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Desmopressin 100µg; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Change From Baseline in Number of Nocturnal Voids After 28 Days of Treatment - Period 2
Description: Records of nocturia and sleep over three consecutive days per week were kept in voiding-sleep diaries by study participants. The average number of nocturnal voids of the 3 days recorded in the last week of the study (between study days 25-32) was compared to average baseline readings.
Time Frame: 3 days between study days -6 to 0 (Baseline), and days 25 to 32
Population: Per protocol population, consisting of treated participants without major protocol violations and with >=80% treatment compliance. Missing values post baseline were imputed using last observation carried forward (LOCF) where at least one post baseline measurement was available at a visit before the missing observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: nocturnal voids
Arm/Group | Placebo | Desmopressin 10µg | Desmopressin 25µg | Desmopressin 50µg | Desmopressin 100µg
Number analyzed (Participants) | 22 | 22 | 20 | 19 | 21
nocturnal voids | -0.735 [-1.049 to -0.421] | -1.007 [-1.320 to -0.695] | -1.282 [-1.583 to -0.981] | -1.589 [-1.903 to -1.274] | -1.624 [-1.999 to -1.248]
Statistical Analysis 1: Comparison: Placebo vs Desmopressin 10µg; Test type: Superiority or Other; p = 0.194, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Gender is a factor, and duration of action and baseline number of nocturnal voids are covariates; Mean Difference (Net) = -0.272, 95% CI 2-sided [-0.685 to -0.141]
Statistical Analysis 2: Comparison: Placebo vs Desmopressin 25µg; Test type: Superiority or Other; p = 0.015, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Gender is a factor, and duration of action and baseline number of nocturnal voids are covariates; Mean Difference (Net) = -0.547, 95% CI 2-sided [-0.985 to -0.108]
Statistical Analysis 3: Comparison: Placebo vs Desmopressin 50µg; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Gender is a factor, and duration of action and baseline number of nocturnal voids are covariates; Mean Difference (Net) = -0.854, 95% CI 2-sided [-1.317 to -0.391]
Statistical Analysis 4: Comparison: Placebo vs Desmopressin 100µg; Test type: Superiority or Other; p = 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Gender is a factor, and duration of action and baseline number of nocturnal voids are covariates; Mean Difference (Net) = -0.888, 95% CI 2-sided [-1.426 to -0.351]

3. Secondary Outcome: Area Under the Urine Osmolality Curve (AUCosm)
Description: Area under the urine osmolality curve, from dose administration to end of action (AUCosm).
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*mOsm/kg
Arm/Group | Placebo | Desmopressin 10µg | Desmopressin 25µg | Desmopressin 50µg | Desmopressin 100µg
Number analyzed (Participants) | 23 | 23 | 22 | 21 | 21
h*mOsm/kg | 0.00 (0.00) | 24.67 (97.50) | 852.00 (1576.10) | 1551.01 (1501.21) | 3112.53 (2131.69)

4. Secondary Outcome: Area Under the Urine Production Curve (AUCurine Prod)
Description: Area under the urine production curve, from dose administration to end of action (AUCurine prod)
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*mL
Arm/Group | Placebo | Desmopressin 10µg | Desmopressin 25µg | Desmopressin 50µg | Desmopressin 100µg
Number analyzed (Participants) | 23 | 23 | 22 | 21 | 23
h*mL | 59.34 (153.78) | 214.24 (266.86) | 297.17 (322.51) | 522.99 (283.90) | 537.08 (330.67)

5. Secondary Outcome: Time When Urine Production <0.12 ml/kg/Min
Description: Urine volume was registered and samples for osmolality check were collected every 30 minutes as long as there was an antidiuretic action defined as a urine production <0.12 mL/kg/min. The hydration due to water-loading should have lasted until end of action, defined as when the urine production returned to >0.12 mL/kg/min, but no longer than 12 hours.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | Desmopressin 10µg | Desmopressin 25µg | Desmopressin 50µg | Desmopressin 100µg
Number analyzed (Participants) | 23 | 23 | 22 | 21 | 23
hours | 0.41 (1.15) | 1.67 (2.16) | 3.50 (4.17) | 6.05 (3.56) | 8.20 (2.59)

6. Secondary Outcome: Change From Baseline in Duration of First Period of Undisturbed Sleep After 28 Days of Treatment - Period 2
Description: Duration of first period of undisturbed sleep is defined as the length of time from initial sleep to first awakening.
  Records of nocturia and sleep over three consecutive days per week were kept in voiding-sleep diaries by study participants. The average length of first period of undisturbed sleep of the 3 days recorded in the last week of the study (between study days 25-32) was compared to average baseline readings.
Time Frame: 3 days between study days -6 to 0 (Baseline), and days 25 to 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Desmopressin 10µg | Desmopressin 25µg | Desmopressin 50µg | Desmopressin 100µg
Number analyzed (Participants) | 22 | 22 | 20 | 19 | 21
minutes | 68.39 (93.32) | 101.85 (120.26) | 113.45 (120.22) | 190.77 (124.32) | 194.25 (99.17)

7. Secondary Outcome: Change From Baseline in Total Sleep Time at Approximately Day 32
Description: Total sleep time is defined as the time spent asleep from initial sleep to final awakening.
  Records of nocturia and sleep over three consecutive days per week were kept in voiding-sleep diaries by study participants. The average of the total time asleep of the 3 days recorded in the last week of the study (between study days 25-32) was compared to average baseline readings.
Time Frame: 3 days between study days -6 to 0 (Baseline), and days 25 to 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Desmopressin 10µg | Desmopressin 25µg | Desmopressin 50µg | Desmopressin 100µg
Number analyzed (Participants) | 22 | 22 | 20 | 19 | 21
minutes | 2.47 (49.94) | -11.86 (48.57) | -33.04 (116.09) | 6.81 (69.04) | 14.07 (54.06)

8. Secondary Outcome: Change From Baseline in Number of Daytime Voids at Approximately Day 32
Description: Number of daytime voids was recorded over three consecutive days per week in diaries kept by study participants. The average number of daytime voids of the 3 days recorded in the last week of the study (between study days 25-32) was compared to the average baseline readings.
Time Frame: 3 days between study days -6 to 0 (Baseline), and days 25 to 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: voids
Arm/Group | Placebo | Desmopressin 10µg | Desmopressin 25µg | Desmopressin 50µg | Desmopressin 100µg
Number analyzed (Participants) | 22 | 22 | 20 | 19 | 21
voids | 0.49 (1.33) | 0.68 (1.53) | 0.15 (1.66) | 0.23 (1.51) | 0.63 (1.74)

9. Secondary Outcome: Change From Baseline in Number of 24-hour Urine Voids at Approximately Day 32
Description: Number of voids in 24 hours was recorded over three consecutive days per week in diaries kept by study participants. The average number of 24-hour voids of the 3 days recorded in the last week of the study (between study days 25-32) was compared to the average baseline readings.
Time Frame: 3 days between study days -6 to 0 (Baseline), and days 25 to 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: voids
Arm/Group | Placebo | Desmopressin 10µg | Desmopressin 25µg | Desmopressin 50µg | Desmopressin 100µg
Number analyzed (Participants) | 22 | 22 | 20 | 19 | 21
voids | -0.15 (1.71) | -0.47 (1.93) | -1.19 (1.85) | -1.33 (1.81) | -0.96 (1.69)

10. Secondary Outcome: Change From Baseline in Nocturnal Urine Volume at Approximately Day 32
Description: Nocturnal urine volume was recorded over three consecutive days per week in diaries kept by study participants. The average nocturnal urine volume of the 3 days recorded in the last week of the study (between study days 25-32) was compared to the average baseline readings.
Time Frame: 3 days between study days -6 to 0 (Baseline), and days 25 to 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Placebo | Desmopressin 10µg | Desmopressin 25µg | Desmopressin 50µg | Desmopressin 100µg
Number analyzed (Participants) | 22 | 22 | 20 | 19 | 21
ml | -114.70 (224.53) | -140.68 (168.62) | -209.87 (262.89) | -295.02 (196.71) | -333.22 (154.05)

11. Secondary Outcome: Change From Baseline in 24-Hour Urine Volume at Approximately Day 32
Description: Twenty-four hour urine volume was recorded over three consecutive days per week in diaries kept by study participants. The average 24-hour urine volume of the 3 days recorded in the last week of the study (between study days 25-32) was compared to the average baseline readings.
Time Frame: 3 days between study days -6 to 0 (Baseline), and days 25 to 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Placebo | Desmopressin 10µg | Desmopressin 25µg | Desmopressin 50µg | Desmopressin 100µg
Number analyzed (Participants) | 22 | 22 | 20 | 19 | 21
ml | -104.47 (386.27) | -19.47 (371.72) | -201.83 (487.49) | -270.53 (344.29) | -187.25 (369.61)

12. Secondary Outcome: Change From Baseline in 24-Hour Urine Production Per Body Weight at Approximately Day 32
Description: Twenty-four hour urine volume was recorded over three consecutive days per week in diaries kept by study participants. Urine volume per body weight was calculated. The average 24-hour urine volume per kg of body weight of the 3 days recorded in the last week of the study (between study days 25-32) was compared to the average baseline readings.
Time Frame: 3 days between study days -6 to 0 (Baseline), and days 25 to 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ml/kg
Arm/Group | Placebo | Desmopressin 10µg | Desmopressin 25µg | Desmopressin 50µg | Desmopressin 100µg
Number analyzed (Participants) | 22 | 22 | 20 | 19 | 21
ml/kg | -2.017 (6.205) | -0.096 (6.814) | -3.523 (7.621) | -4.573 (6.183) | -3.058 (6.263)

13. Secondary Outcome: Change From Baseline in Nocturnal Polyuria Index at Approximately Day 32
Description: Nocturnal polyuria index is defined as a proportion of nocturnal urine volume to the 24-hour urine volume. Urine volume and time of day of those voids was recorded over three consecutive days per week in diaries kept by study participants. The average nocturnal polyuria index of the 3 days recorded in the last week of the study (between study days 25-32) was compared to the average baseline readings.
Time Frame: 3 days between study days -6 to 0 (Baseline), and days 25 to 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nocturnal urine volume / 24-hour urine
Arm/Group | Placebo | Desmopressin 10µg | Desmopressin 25µg | Desmopressin 50µg | Desmopressin 100µg
Number analyzed (Participants) | 22 | 22 | 20 | 19 | 21
nocturnal urine volume / 24-hour urine | -4.72 (6.75) | -7.82 (6.65) | -8.61 (9.28) | -13.56 (9.72) | -16.00 (6.87)

14. Secondary Outcome: Change From Baseline in Nocturia-Related Quality of Life Based on Evaluation Provided by Nocturia Quality of Life Questionnaire (N-QoL) at Approximately Day 32
Description: N-QoL assesses the impact of nocturia on quality of life (QoL) and treatment outcomes. N-QoL is a self-administered questionnaire with 13 items using scales of 0 = no negative impact to QoL to the upper number = signficant negative impact to QoL. The sleep/energy domain consists of 7 questions with a scale of 0 to 28. The bother/concern domain consists of 5 questions for a scale of 0 to 20. The 13th question is an overall assessment scored from 0 to 10. The Total Score includes all 13 questions with a scale of 0 (no negative impact to QoL) to 58 (significant negative impact to QoL).
Time Frame: Approximately Day 4 (start of period 2) and Day 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Desmopressin 10µg | Desmopressin 25µg | Desmopressin 50µg | Desmopressin 100µg
Number analyzed (Participants) | 22 | 23 | 22 | 21 | 22
units on a scale
  Sleep/Energy subscale | 7.77 (11.66) | 10.69 (15.33) | 13.26 (15.46) | 12.30 (10.82) | 8.52 (12.23)
  Bother/Concern subscale | 6.36 (19.02) | 8.99 (16.91) | 16.33 (18.35) | 10.67 (19.37) | 10.15 (14.00)
  Total Score | 7.04 (14.05) | 9.98 (14.65) | 14.78 (16.28) | 11.44 (13.00) | 9.39 (11.11)

15. Secondary Outcome: Change From Baseline in Sleep Related Quality of Life Based on the Global Score of the Pittsburgh Sleep Quality Index (PSQI) at Approximately Day 32
Description: The Global Score of the Pittsburgh Sleep Quality Index (PSQI) is comprised of Questions 2-9 with a total scale of 0 (no difficulty sleeping) to 21 (severe difficulty). The change in Global Score is Global Score at the end of period 2 (day 32) - Global Score at the start of Period 2 (day 4). A negative change indicates an improvement in quality of life.
Time Frame: Approximately Day 4 (start of period 2) and Day 32
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Desmopressin 10µg | Desmopressin 25µg | Desmopressin 50µg | Desmopressin 100µg
Number analyzed (Participants) | 22 | 23 | 21 | 21 | 21
units on a scale | -1.2 (2.0) | -0.6 (2.3) | -1.5 (2.2) | -1.4 (2.5) | -1.3 (1.8)

16. Secondary Outcome: Participant Counts of Minimum Observed Serum Sodium Levels During the Second Treatment Period (Days 4-32)
Description: Serum sodium levels were monitored throughout the trial as part of the clinical chemistry panel. If the value was ≤125 mEq/L, the participant was to be withdrawn from the trial and treatment stopped immediately. This outcome reports participants' lowest recorded serum sodium levels during the second treatment period.
Time Frame: Days 4- 32
Population: Safety population which included all randomised and exposed participants. Participants were analysed according to the actual treatment received.
Measure: Number; unit: participants
Arm/Group | Placebo | Desmopressin 10µg | Desmopressin 25µg | Desmopressin 50µg | Desmopressin 100µg
Number analyzed (Participants) | 23 | 23 | 22 | 22 | 23
participants
  >= 135 mEq/L | 23 | 23 | 21 | 21 | 23
  >=130 mEq/L to <135 mEq/L | 0 | 0 | 1 | 1 | 0
  <130 mEq/L | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Period 1: Day 1 to Day 3 (includes Wash-out period) Period 2: Day 4 (first day of period 2 drug administration) to Day 32 (last day of drug administration or date of withdrawal)
Groups:
- Placebo-Period 1: Study period 1: single dose of placebo.
- Desmopressin 10µg - Period 1: Study period 1: single dose of desmopressin 10µg.
- Desmopressin 25µg - Period 1: Study period 1: single dose of desmopressin 25µg.
- Desmopressin 50µg - Period 1: Study period 1: single dose of desmopressin 50µg.
- Desmopressin 100µg - Period 1: Study period 1: single dose of desmopressin 100µg.
- Placebo - Period 2: Study period 2: daily doses of placebo taken before bedtime for 28 days.
- Desmopressin 10µg - Period 2: Study period 2: daily doses of desmopressin 10µg taken before bedtime for 28 days.
- Desmopressin 25µg - Period 2: Study period 2: daily doses of desmopressin 25µg taken before bedtime for 28 days.
- Desmopressin 50µg - Period 2: Study period 2: daily doses of desmopressin 50µg taken before bedtime for 28 days.
- Desmopressin 100µg - Period 2: Study period 2: daily doses of desmopressin 100µg taken before bedtime for 28 days.
Arm/Group | Placebo-Period 1 | Desmopressin 10µg - Period 1 | Desmopressin 25µg - Period 1 | Desmopressin 50µg - Period 1 | Desmopressin 100µg - Period 1 | Placebo - Period 2 | Desmopressin 10µg - Period 2 | Desmopressin 25µg - Period 2 | Desmopressin 50µg - Period 2 | Desmopressin 100µg - Period 2
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/25 | 0/22 | 0/22 | 0/24 | 0/23 | 0/23 | 0/22 | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 1/25 | 1/22 | 4/22 | 7/24 | 3/23 | 1/23 | 4/22 | 1/22 | 0/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-Period 1 (N=23) | Desmopressin 10µg - Period 1 (N=25) | Desmopressin 25µg - Period 1 (N=22) | Desmopressin 50µg - Period 1 (N=22) | Desmopressin 100µg - Period 1 (N=24) | Placebo - Period 2 (N=23) | Desmopressin 10µg - Period 2 (N=23) | Desmopressin 25µg - Period 2 (N=22) | Desmopressin 50µg - Period 2 (N=22) | Desmopressin 100µg - Period 2 (N=23)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.